CLINICAL TRIAL: NCT05773950
Title: Comparison of Dual Therapy of Dexamethasone and Palonosetron and Triple Therapy of Dexamethasone, Palonosetron, Fosaprepitant for Postoperative Nausea and Vomiting Prevention: a Randomized Controlled Trial
Brief Title: Triple Therapy of Dexamethasone, Palonosetron, and Fosaprepitant As PONV Prevention
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Heejoon Jeong, Assistant professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SMC2022-12-050-001
Record Dates: First submitted 2023-03-07; First posted 2023-03-17 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-01

CONDITIONS: Postoperative Nausea and Vomiting; Gynecologic Surgical Procedures; Laparoscopy
Keywords: PONV; fosaprepitant; dexamethasone; palonosetron
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — fosaprepitant; Aprepitant; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dual therapy group (Placebo Comparator): On the day of surgery, in the preoperative holding area, the principal investigator administers the study drug to the participants. During the study drug administration period, the principal investigator observes the presence of specific symptoms and abnormalities at the injection site of participants.
  In the case of the control group, the study drug is 150 ml of normal saline, which is visually indistinguishable from the dilute solution of the fosaprepitant, administered over 30 minutes.
  The subject is then moved to the operating room and undergoes induction of general anesthesia. After the induction of anesthesia, 5 mg of dexamethasone and 0.075 mg of palonosetron are intravenously administered.
  Interventions: Drug: normal saline
- Triple therapy group (Experimental): On the day of surgery, in the preoperative holding area, the principal investigator administers the study drug to the participants. During the study drug administration period, the principal investigator observes the presence of specific symptoms and abnormalities at the injection site of participants. In the case of the experimental group, 150 ml of normal saline mixed with 150 mg of fosaprepitant is administered over 30 minutes.
  The subject is then moved to the operating room and undergoes induction of general anesthesia. After the induction of anesthesia, 5 mg of dexamethasone and 0.075 mg of palonosetron are intravenously administered.
  Interventions: Drug: fosaprepitant

INTERVENTIONS:
Drug: fosaprepitant — The subject is then moved to the operating room and undergoes induction of general anesthesia. After the induction of anesthesia, 5 mg of dexamethasone and 0.075 mg of palonosetron are intravenously administered.
  In the experimental group, the subject is then moved to the operating room and undergoes induction of general anesthesia. After the induction of anesthesia, 5 mg of dexamethasone and 0.075 mg of palonosetron are intravenously administered.
  Other Names: emend
  Arms: Triple therapy group
Drug: normal saline — On the day of surgery, in the preoperative holding area, the principal investigator administers the study drug to the participants. During the study drug administration period, the principal investigator observes the presence of specific symptoms and abnormalities at the injection site of participants.
  In the case of the control group, the study drug is 150 ml of normal saline, which is visually indistinguishable from the dilute solution of the fosaprepitant, administered over 30 minutes.
  Other Names: placebo
  Arms: Dual therapy group

SUMMARY:
As a preventive for postoperative nausea and vomiting in patients undergoing laparoscopic gynecological surgery, the investigators shall investigate the efficacy of the triple therapy of dexamethasone, palonosetron, and fosaprepitant comparing to dual therapy of dexamethasone and palonosetron.

DETAILED DESCRIPTION:
Intervention

1. Control group (dual therapy) study drug (placebo): normal saline 150ml Dexamethasone 5 mg palonosetron 0.075 mg,
2. Experimental group (triple therapy) Study Drug (Fosaprepitant): resolved in normal saline 150mL Dexamethasone, Palonosetron 0.075mg,

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic gynecological surgery.
* Adults between the ages of 18 and 50
* American Society of Anesthesiologists Physical Status (ASA physical status I, II

Exclusion Criteria:

* American Association of Anesthesiologists physical standards (ASA physical status III or higher)
* Children under the age of 19
* Adults over 49 years of age
* Diabetes Mellitus
* Pregnant or lactating women
* Patients with a history of allergy or contraindications for use of the study drug
* Patients who did not understand this study or expressed their refusal.
* Patients with a history of serious psychologic disease that may affect the patient evaluation
* Patients taking serotonergic drugs

Ages: 19 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
the incidence of Postoperative nausea and vomiting | during 24 hours after surgery
  yes or no

SECONDARY OUTCOMES:
the incidence of Postoperative nausea and vomiting | during post-anesthesia care unit stay, during 6 hours after surgery
  yes or no
the severity of Postoperative nausea and vomiting | during post-anesthesia care unit stay, during 6 hours after surgery, during 24 hours after surgery
  numeric rating scale 0-10 and PONV impact scale
rescue antiemetics | during 24 hours after surgery
  dose
time to rescue antiemetics | during 24 hours after surgery
  the first administration time point of rescue antiemetics
postoperative pain at rest and couging | during post-anesthesia care unit stay, during 6 hours after surgery, during 24 hours after surgery
  numeric rating scale 0-10
opioid consumption | during 24 hours after surgery
  morphine equivalent dose
Any adverse event | during 24 hours after surgery
  yes or no
Time to normal diet | during 24 hours after surgery
  time of succes of normal diet
Qualityof recovery from surgery and anesthesia | during 24 hours after surgery
  QoR 15K questionairre
Time to first flatus | during in hospital stay, an average of 5 days
  gas out time pointsyes or no

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea